CLINICAL TRIAL: NCT02915861
Title: Eschar Investigations to Improve Diagnostics, Understand Early Immune Responses and Characterize Strains for Vaccines in Scrub Typhus
Brief Title: Eschar Investigations in Scrub Typhus
Acronym: EXIST
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Chiangrai Prachanukroh Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO1504
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Scrub Typhus
Keywords: immune responses; vaccines
MeSH Terms: conditions — Scrub Typhus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Non-invasive eschar samples
  2. Eschar biopsy
  3. Lymph node fine-needle aspiration biopsy (LN FNA)
  4. Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- EXPa: Scrub typhus patients: Group A
  Interventions: Other: Non-invasive eschar samples + blood
- EXPb: Scrub typhus patients: Group B
  Interventions: Other: Non-invasive eschar samples+eschar biopsy+blood
- EXPc: Scrub typhus patients: Group C
  Interventions: Other: Non-invasive eschar samples+eschar biopsy+lymph node fine-needle aspiration biopsy+blood
- EXC: Control group
  Interventions: Other: Blood+Skin sample

INTERVENTIONS:
Other: Non-invasive eschar samples + blood — EXPa (n=12) will have blood and non-invasive eschar samples collected (consent to study, declined biopsy).
  Groups: EXPa
Other: Non-invasive eschar samples+eschar biopsy+blood — EXPb (n=12) will have blood, non-invasive eschar samples, and an eschar biopsy collected (consent to study, draining LN inaccessible).
  Groups: EXPb
Other: Non-invasive eschar samples+eschar biopsy+lymph node fine-needle aspiration biopsy+blood — EXPc (n=12) will have blood, non-invasive eschar samples, eschar biopsy, and LN FNA collected (consent to study, draining LN accessible).
  Groups: EXPc
Other: Blood+Skin sample — Controls (EXC, n=12) are healthy individuals, attending hospital for elective/minor surgery or treatment of minor skin injury, and normally reside in a scrub typhus endemic region. Blood and a skin sample will be collected at baseline only.
  Groups: EXC

SUMMARY:
This is an observational study of patients with scrub typhus (rapid diagnostic test/quantitative polymerase chain reaction (RDT/qPCR) positive) and an inoculation eschar present on examination, recruited from Chiangrai Prachanukroh Hospital, North of Thailand.

In this study, we aim to:

* Investigate relevant pathogen dissemination dynamics, early innate immune response, and pathogen-host interactions in scrub typhus using a minimal set of easily accessible samples; the inoculation eschar (crust or biopsy), whole blood and - where possible - a lymph node fine-needle aspiration (FNA).
* Determine the potential use of the inoculation eschar for improving early diagnostics and assessing the diversity of human pathogenic strains; by evaluating non-invasive swabs and scrapings, as well as biopsies for molecular diagnostics templates.
* Dissect the underlying patho-biology associated with the inoculation eschar and in a subgroup, including the draining lymph node; by defining the spectrum of infected cells via microscopy and double-immune labeling; by determining cytokine and RNA gene expression profiles in blood peripheral blood mononuclear cell (PBMCs) and eschar samples.

Data sharing:

No future analysis or study of legacy data/specimens including data sharing for purposes not specified in the protocol will be done without seeking further regulatory (EC/IRB) approval

* Any requests for data sharing will be considered by MORU's data sharing committee
* Any data subsequently shared will be anonymised and will not include personal identifiers

DETAILED DESCRIPTION:
Scrub typhus patients will be recruited into the scrub typhus patient (EXP) arm of the study. There will be 3 sub-groups:

* EXPa (n=12) will have blood and non-invasive eschar samples collected (consent to study, declined biopsy).
* EXPb (n=12) will have blood, non-invasive eschar samples, and an eschar biopsy collected (consent to study, draining lymph node (LN) inaccessible).
* EXPc (n=12) will have blood, non-invasive eschar samples, eschar biopsy, and LN FNA collected (consent to study, draining LN accessible).

Samples will be collected at baseline (all) and 2 weeks (blood only).

Control participants will be recruited into the scrub typhus control.

- EXC (n=12) are healthy individuals, attending hospital for elective/minor surgery or treatment of minor skin injury, and normally reside in a scrub typhus endemic region. Blood and a skin sample will be collected at baseline only.

ELIGIBILITY:
Scrub Typhus Patients (EXP) inclusion criteria:

* Age ≥7 years old.
* Presentation to hospital with fever in ≤14 days and a clinical suspicion of typhus.
* Eschar observed on examination.
* Scrub typhus RDT positive or OT qPCR positive (if qPCR available at local site by time of study initiation).
* Willingness to participate in the study. Written informed consent obtained from the patient (≥18 years old) or, written informed assent from participant (≥7 to <18years old) along with written informed consent from participant's parent(s)/legal guardian(s).

Scrub Typhus Controls (EXC) inclusion criteria:

* Age ≥7 years old.
* Clinically well, attending elective/minor surgery or for treatment of minor skin injury.
* Historical diagnosis of scrub typhus (RDT, serology, and/or PCR positivity) more than 2 years ago or living in an endemic area with high risk of previous exposure.
* Willingness to participate in the study. Written informed consent obtained from the patient (≥18 years old) or written informed assent from participant (≥7 to <18years old) along with written informed consent from participant's parent(s)/legal guardian(s).

Scrub Typhus Patients (EXP) exclusion criteria:

* Current TB or TB treatment in ≤6 months (contains OT-effective antimicrobials)
* Documented HIV infection, use of steroids, chemotherapy, other immunosuppressants, or herbal remedies containing steroids, and/or pregnancy

Scrub Typhus Controls (EXC) exclusion criteria:

* Significant acute intercurrent illness at the time of admission including fever >37.5˚C or infection (including TB) requiring antibiotics
* Documented HIV infection, use of steroids, chemotherapy, other immunosuppressants, or herbal remedies containing steroids, and/or pregnancy

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EXP: Male and female patients ≥7 years old with confirmed acute scrub typhus and an eschar present on examination (N=36).
  EXC: Healthy individuals ≥7 years old who normally reside in a scrub typhus endemic region, attending hospital for elective/minor surgery or treatment of minor skin injury, and preferably age and sex-matched (N=12).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Phenotypic characterisation of the major subset of Orientia tsutsugamushi (OT) infected leucocytes within eschar, lymph node, and blood during the dissemination phase of OT in vivo. | 2 years
Characterisation of cytokine and RNA gene expression profiles within the eschar, lymph node, and blood in vivo and comparisons with profiles of uninfected target cells. | 2 years

SECONDARY OUTCOMES:
Establishing the usefulness of non-invasive eschar samples from patients with acute scrub typhus for diagnostics for OT and for genotyping +/- whole-genome sequencing. | 2 years
Define and contrast the eschar histo-pathological findings in this study in Thailand to previous findings from Laos, where the Gilliam strain predominates. | 2 years
Comparisons to parallel studies in the non-human primate model with emphasis on dissemination dynamics, immunomodulation, and the innate and adaptive immune responses to OT; contributing to vaccine development. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tri Wangrangsimakul, MD, Principal Investigator — Chiangrai Prachanukroh Hospital, Chiangrai, Thailand
Locations (1):
- Chiangrai Prachanukroh Hospital, Chiang Rai, Thailand

IPD SHARING:
Plan to Share IPD: No